CLINICAL TRIAL: NCT00344877
Title: Anticonvulsive Effects of Transcranial DC Stimulation in Pharmacoresistant Focal Epilepsy
Brief Title: Electrical Brain Stimulation to Reduce Epileptic Seizures
Status: Completed | Type: Observational
Sponsor: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 060187; 06-N-0187
Record Dates: First submitted 2006-06-23; First posted 2006-06-27 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2009-05-05

CONDITIONS: Temporal Lobe Epilepsy
Keywords: Epilepsy; Temporal Lobe Epilepsy; Cortical Excitability; Transcranial Direct Current Stimulation (tDCS); Memory Testing; Seizures; Transcranial Magnetic Stimulation (TMS); Memory; Plasticity
MeSH Terms: conditions — Epilepsy, Temporal Lobe; Epilepsy; Seizures

SUMMARY:
OBJECTIVES:

About 15% of patients suffering from focal epilepsy are refractory to available pharmacological treatments. Until now, the only hope for such patients has been the development of new pharmaceutical treatments or epilepsy surgery. In case of inoperability, different types of invasive brain stimulation such as vagus nerve stimulation or deep brain stimulation or non-invasive repetitive TMS have been evaluated to determine their anticonvulsive potential. For rTMS, weak and short lasting seizure reduction has been reported in different epilepsy syndromes.

A new, non-invasive stimulation technique, transcranial direct current stimulation (tDCS), was useful to modulate cortical excitability in many cortical areas (M1, visual cortex, frontal cortex). Cathodal tDCS, with a current of 1 mA, induced long-term depression in animal models and reportedly decreased the excitability of both human and animal cerebral cortex. In epilepsy patients suffering from a malformation of cortical development, a single session of cathodal tDCS helped reduce seizures briefly. The purpose of this protocol is to study the effects of repeated applications of tDCS on the excitability of the seizure focus in patients with poorly controlled pharmacologically refractory temporal lobe epilepsy.

STUDY POPULATION:

We plan to study 56 patients between the ages of 18 and 80 suffering from temporal lobe epilepsy.

DESIGN:

Subjects will be allocated by blocked randomization to one of two groups (parallel design). Group A will receive cathodal tDCS and group B will receive Sham-tDCS on five consecutive days. Each subject will participate in 9 sessions (1 baseline visit, 5 intervention visits, 3 follow-up visits). The effect of the intervention relative to the sham stimulation will be evaluated by comparing seizure frequency and neuropsychological tests during the 8 weeks before and after the intervention.

OUTCOME MEASURES:

Primary outcome measure will be the mean seizure frequency per 4 weeks in the tDCS group as compared to the Sham-tDCS group. To analyze the effect of the intervention (tDCS), seizures will be evaluated during a 2x4 week baseline period before tDCS and 2x4 weeks after the intervention. Using these data we will calculate the percentage change of seizures per 4 weeks.

Secondary outcome measures will be the scores of the neuropsychological testing (HVLT-R, BVMT-R, CTMT, COWAT) and number of epileptiform discharges in the EEG. Furthermore, th...

DETAILED DESCRIPTION:
OBJECTIVES:

About 15% of patients suffering from focal epilepsy are refractory to available pharmacological treatments. Until now, the only hope for such patients has been the development of new pharmaceutical treatments or epilepsy surgery. In case of inoperability, different types of invasive brain stimulation such as vagus nerve stimulation or deep brain stimulation or non-invasive repetitive TMS have been evaluated to determine their anticonvulsive potential. For rTMS, weak and short lasting seizure reduction has been reported in different epilepsy syndromes.

A new, non-invasive stimulation technique, transcranial direct current stimulation (tDCS), was useful to modulate cortical excitability in many cortical areas (M1, visual cortex, frontal cortex). Cathodal tDCS, with a current of 1 mA, induced long-term depression in animal models and reportedly decreased the excitability of both human and animal cerebral cortex. In epilepsy patients suffering from a malformation of cortical development, a single session of cathodal tDCS applied to various cortical areas including frontal and temporal cortex helped reduce seizures briefly. The purpose of this protocol is to study the effects of repeated applications of tDCS on the excitability of the seizure focus in patients with poorly controlled pharmacologically refractory frontal and/or temporal lobe epilepsy.

STUDY POPULATION:

We plan to study 56 patients between the ages of 18 and 80 suffering from frontal and/or temporal lobe epilepsy.

DESIGN:

Subjects will be allocated by blocked randomization to one of two groups (parallel design). Group A will receive cathodal tDCS and group B will receive Sham-tDCS on five consecutive days. Each subject will participate in 9 sessions (1 baseline visit, 5 intervention visits, 3 follow-up visits). The effect of the intervention relative to the sham stimulation will be evaluated by comparing seizure frequency and neuropsychological tests during the 8 weeks before and after the intervention.

OUTCOME MEASURES:

Primary outcome measure will be the mean seizure frequency per 4 weeks in the tCDS group as compared to the Sham-tDCS group. To analyze the effect of the intervention (tDCS), seizures will be evaluated during a 2x4 week baseline period before tDCS and a 2x4 weeks after the intervention. Using these data we will calculate the percentage change of seizures/4 weeks.

Secondary outcome measures will be the scores of the neuropsychological testing (HVLT-R, BVMT-R, CTMT, COWAT) and number of epileptiform discharges in the EEG. Furthermore, the patients will answer several questionnaires to evaluate quality of life (QOLIE-31-P), seizure severity (SSQ), and mood (BDI). To better understand the mechanisms underlying the proposed change of seizure frequency, we will use single- and paired- pulse transcranial magnetic stimulation (TMS) to identify corticomotor excitability changes.

ELIGIBILITY:
* INCLUSION CRITERIA:

Patients will be included under the following circumstances:

1. Age between 18 to 80 years.
2. Written informed consent is given by the patient.
3. Epileptogenic focus in the temporal lobe or in the frontal lobe (unilateral or bilateral with dominant focus).
4. Seizures are not completely responsive to medical treatment (8 or more seizures per month for at least 3 months) and patients have failed at least two anticonvulsant regimens in the past. The implantation of a vagus nerve stimulator will also be counted as anticonvulsant regimen.
5. A stable anticonvulsant regimen (not more than three anticonvulsants) defined as unchanged dose or dose modifications lower than 20% in the last month (Blood levels of anticonvulsants will be measured at the beginning of the study, prior and after intervention, and after the study to assure that the type and dose of medication remains constant). For the vagus nerve stimulator, the stimulation parameters will have to be unchanged for at least one month.
6. One antidepressant on a stable dose regimen for at least 1 month will be allowed.
7. Mini-Mental-Status examination greater than or equal to 23 points.
8. Commitment to participate in the long-term follow-up (up to 5 months).

EXCLUSION CRITERIA:

We will exclude patients if one of the following conditions applies:

1. A history of any neurological illness other than the epilepsy.
2. Acute symptomatic seizures (caused by brain tumor, acute stroke, intracranial hemorrhage, encephalitis) or psychogenic seizures.
3. Generalized epilepsy or focal epilepsy with the epileptogenic zone outside the temporal lobe.
4. A history of severe alcohol or drug abuse; psychiatric illness such as severe, clinically significant depression (as evaluated by BDI); poor motivational capacity; or severe language disturbances, particularly of receptive nature or with serious cognitive deficits.
5. More than moderate uncontrolled medical problems (e.g., cardiovascular disease, active cancer or renal disease, any kind of end-stage pulmonary or cardiovascular disease, hypo/hyperthyroidism, severe diabetes, peripheral arteriopathy, or a deteriorated condition due to age, or other medical conditions as determined by the study physician, that would interfere with participation in this study).
6. Increased intracranial pressure as evaluated by clinical means (presence of papilledema in eye ground exam, compressed sulci/ventricle on MRI scan).
7. Previous implantation of metallic material (e.g., vascular clips, cochlear implant) in the cranium (except in the mouth), pacemaker, implanted medication pumps, neural stimulators. This does not apply for implantation of a vagus nerve stimulator (Cyberonics ® (Registered Trademark) [Registered Trademark] 100, 102 or 102R).
8. Drug treatment acting primarily on the central nervous system (other than the regular anticonvulsant treatment and one antidepressant) that lowers the seizure threshold such as antipsychotic drugs (chlorpromazine, clozapine) or tricyclic antidepressants.
9. Diseased or damaged skin over the face or scalp.
10. Pregnancy.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56
Dates: Start 2006-06-19; Study Completion 2009-05-05

CONTACTS AND LOCATIONS:
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Sander JW. Some aspects of prognosis in the epilepsies: a review. Epilepsia. 1993 Nov-Dec;34(6):1007-16. doi: 10.1111/j.1528-1157.1993.tb02126.x. PMID 8243349
- [Background] Sander JW, Shorvon SD. Epidemiology of the epilepsies. J Neurol Neurosurg Psychiatry. 1996 Nov;61(5):433-43. doi: 10.1136/jnnp.61.5.433. No abstract available. PMID 8965090
- [Background] Theodore WH, Hunter K, Chen R, Vega-Bermudez F, Boroojerdi B, Reeves-Tyer P, Werhahn K, Kelley KR, Cohen L. Transcranial magnetic stimulation for the treatment of seizures: a controlled study. Neurology. 2002 Aug 27;59(4):560-2. doi: 10.1212/wnl.59.4.560. PMID 12196649